CLINICAL TRIAL: NCT04205799
Title: A Phase II Study Assessing Safety and Efficacy of Cabozantinib for Advanced or Metastatic Cervical Carcinoma After Platinum Treatment Failure
Brief Title: Cabozantinib for Advanced or Metastatic Cervical Carcinoma After Platinum Treatment Failure
Acronym: CABOCOL-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002184-97
Record Dates: First submitted 2019-11-28; First posted 2019-12-19 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Advanced/Metastatic Cervical Cancer
Keywords: cervical cancer; advanced/metastatic; Cabozantinib; platinum treatment failure
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CABOZANTINIB (Experimental): Cabozantinib will be administered at the daily dose of 60 mg given orally in a 4-week cycle. It will be continued without interruption until disease progression or discontinuation for any cause.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib will be administered at the daily dose of 60 mg given orally in a 4-week cycle. It will be continued without interruption until disease progression or discontinuation for any cause.

SUMMARY:
Assess efficacy and safety of cabozantinib in monotherapy in advanced/metastatic cervical cancer (CC) after failure of platinum-based regimen treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years of age or older
* Histologically confirmed recurrent unresectable or metastatic cervix carcinoma with squamous cell, adenocarcinoma or adenosquamous histology - - Patient may have received at least one prior chemotherapy regimen of platinum-based chemotherapy for recurrence or metastatic disease.
* Cisplatin given in combination with radiation for a localized disease does not count as a prior chemotherapy.
* Prior treatment for advanced/metastatic disease with bevacizumab is allowed.
* Prior treatments with immune checkpoint inhibitors are allowed. - ECOG performance status 0-2 - Measurable disease per RECIST 1.1
* The subject must have recovered to baseline or CTCAE v.5.0 (Common Terminology Criteria for Adverse Events, version 5.0) ≤ Grade 1 from clinical toxicities related to any prior treatments, i.e chemotherapy or pelvis radiation unless AE(s) are clinically non-significant (for example alopecia)
* Adequate organ and marrow function, defined as follows, based upon laboratory tests performed within 7 days before inclusion:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3 (≥ 1.0 GI/L)
  * Platelets ≥ 100,000/mm3 (≥ 100 GI/L)
  * Hemoglobin ≥ 10 g/dL (≥ 100 g/L) (red blood cell transfusion is allowed)
  * Total bilirubin ≤ 1.5 fold the upper limit of normal (for subjects with Gilbert's disease, ≤ 3 mg/dL or ≤ 51.3 μmol/L) o Serum albumin ≥ 3.0 g/dL (≥ 30 g/L)
  * Calculated creatinine clearance ≥ 30 mL/min by the CKD-EPI method.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 x the upper limit of normal
  * Urine protein/creatinine ratio (UPCR) ≤ 1g/g (≤ 113.17 mg/mmol creatinine) or 24-hour urine protein < 1 g
* Left-ventricular ejection fraction ≥ 50%
* Subjects affiliated to an appropriate social security system
* Female subjects of childbearing potential must not be pregnant at screening and during treatment by Cabozantinib. Effective methods of contraception should be used throughout the course of treatment and for at least 4 months after the end of treatment. Sexually active fertile subjects and their partners must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the study and 4 months after the last dose of study treatment, even if oral contraceptives are also used.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding and/or fistula / perforation including, but not limited to: Active peptic ulcer disease, inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), history of abdomino and/or pelvic fistula, gastrointestinal perforation, or intra-abdominal abscess, gastro-intestinal obstruction
* Patients with lesions on baseline pelvic MRI which may major the risk of abdominal and/or pelvic fistula/perforation
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations (Note: patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not take cabozantinib and are also excluded).
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA), serious cardiac arrythmias.
* Corrected QT interval (QTc) calculated by the Fridericia formula > 500 msec within 28 days before inclusion (see Annex for Fridericia formula). Note: if initial QTcF is found to be > 500 msec, two additional ECGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 500 msec, the subject meets eligibility in this regard.
* Uncontrolled hypertension defined as systolic blood pressure (SBP) of > 150 mmHg or diastolic blood pressure (DBP) of > 100 mmHg despite an optimal treatment.
* History of cerebrovascular accident including transient ischemic attack (TIA), symptomatic pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT or asymptomatic pulmonary embolism who have been treated with therapeutic anti-coagulating agents for at least 4 weeks are eligible.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or pathologic conditions that carry high risk of bleeding such as coagulopathy or tumor involving major vessels.
* At least 6 weeks must have elapsed between the last dose of pelvis palliative radiation and the first dose of cabozantinib or 2 weeks for other localization of palliative radiation
* Presence of brain metastases or epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before inclusion. Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of inclusion.
* Concomitant use of known strong CYP3A4 inhibitors or inducers.
* Patients with second primary cancer, except adequately treated non-melanoma skin cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 3 years
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Concurrent participation in any therapeutic clinical trial
* Patient deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
efficacy of cabozantinib: proportion of patients with disease control rate | 3 months after cabozantinib treatment initiation.
  Efficacy assessed by the proportion of patients with disease control rate
Safety of cabozantinib: proportion of patients with clinical gastro-intestinal (GI) perforation/fistula, GI-vaginal fistula and genito-urinary (GU) fistula events grade ≥ 2 (NCI CTCAE v 5.0) | toxicities occurring up to 1 month after the end of treatment
  Safety assessed by the proportion of patients with clinical gastro-intestinal (GI) perforation/fistula, GI-vaginal fistula and genito-urinary (GU) fistula events grade ≥ 2 (NCI CTCAE v 5.0)

SECONDARY OUTCOMES:
Objective response (RECIST v1.1 criteria) | At the end of cycle 3,6,9... (each cycle is 28 days) through study completion, an average of 1 year
  Objective response rate defined as the percentage of patients who have achieved complete response or partial response with RECIST 1.1 criteria.
Progression-free survival (PFS) | At the end of cycle 3,6,9... (each cycle is 28 days) through study completion, an average of 1 follow-up year
  Progression-free survival, defined as the time between initiation of cabozantinib treatment and progression (RECIST 1.1 criteria) or death of any cause whichever occurs first.
Overall survival | through study completion, an average of 1 follow-up year
  Overall survival, defined as the time between initiation of cabozantinib treatment and death of whatever cause.
Safety profile of cabozantinib | every cycle of treatment (each cycle is 28 days) through study completion, an average of 1 follow-up year
  Toxicities evaluated according to NCI CTCAE v5.0 criteria, in terms of kind, grade, time of onset, reversibility
Incidence of treatment Quality-of-life of patients assessed by EORTC QLQ-C30 /CX24 questionnaire | At Day 15 of cycle 2 (each cycle is 28 days) and every 3 cycles of treatment ((every 12 weeks)) an average of 1 follow-up year
  Scores of Quality-of-life according to French versions of the self-administered standardized validated questionnaire: EORTC QLQ-C30 with CX24

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Institut de cancérologie de l'Ouest, Angers
  - Centre François Baclesse, Caen
  - Centre Oscar LAMBRET, Lille
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Montpellier, Montpellier
  - Institut de cancérologie de l'Ouest, Nantes
  - Institut CURIE, Saint-Cloud
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coquan E, Brachet PE, Licaj I, Leconte A, Castera M, Lequesne J, Meriaux E, Bonnet I, Lelaidier A, Clarisse B, Joly F. CABOCOL-01 trial: a single-arm phase II study assessing safety and efficacy of Cabozantinib for advanced or metastatic cervical carcinoma after platinum treatment failure. BMC Cancer. 2021 Sep 25;21(1):1054. doi: 10.1186/s12885-021-08758-9. PMID 34563169